CLINICAL TRIAL: NCT05372848
Title: Clinical Evaluation of an Electric and a Manual Toothbrush in Removal of Dental Plaque by Intraoral Imaging Systems
Brief Title: Clinical Evaluation of an Electric and a Manual Toothbrush in Removal of Dental Plaque
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: mudis34
Record Dates: First submitted 2022-05-06; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Plaque, Dental
Keywords: manual toothbrush; electric toothbrush; fluorescence; intraoral scanner; FluoreCam
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Group 1 includes volunteers who used to use manual toothbrushes and started to use an electric toothbrush for 1 month with the same daily brushing routine. Fifteen healthy individuals between the ages of 20 and 30 years with no systemic disease, restoration or caries, and whom have the criteria for using a manual toothbrush for at least 2 years included in Group 1.
  Interventions: Diagnostic Test: Manual toothbrush
- Group 2 (Other): Group 2 includes volunteers who used to use an electric toothbrush and started to use a manual toothbrush for 1 month with the same daily brushing routines. Fifteen healthy individuals between the ages of 20 and 30 years with no systemic disease, restoration or caries, and whom have the criteria for using an electric toothbrush for at least 2 years included in Group 2.
  Interventions: Diagnostic Test: Electric toothbrush

INTERVENTIONS:
Diagnostic Test: Manual toothbrush — volunteers who used manual toothbrush for at least 2 years
  Arms: Group 1
Diagnostic Test: Electric toothbrush — volunteers who used electric toothbrush for at least 2 years
  Arms: Group 2

SUMMARY:
The study aimed to evaluate the efficacy of manual and electric toothbrush on dental plaque removal by using various intraoral imaging systems. Thirty healthy individuals using the same type of toothbrush for at least 2 years participated in the study. 12 teeth of each individual, including upper and lower anteriors, were examined. Group 1 including volunteers who used to use manual toothbrushes (MT) started to use an electric toothbrush (ET) and Group 2 including volunteers who used to use an ET and started to use a MT for 1 month with the same daily brushing routines. Following the clinical intraoral examination, plaque (PI) and gingival index (GI) measurements were performed 5 hours after brushing. The GI was evaluated through Sillness&Löe Gingival Index. The PI was evaluated according to Quigley and Hein's Plaque Index criteria and was scored clinically on visual inspection and digital imaging systems including FluoreCam, DSLR Camera, D-Light Pro, Smile Lite MDP, iTero Element Flex. The data was evaluated under p<0.005 significant level.

DETAILED DESCRIPTION:
Patient and teeth selection criteria Ten healthy individuals between the ages of 20 and 30 years with no systemic disease, restoration or caries, and whom have the criteria for using the same type of toothbrush for 2 years (15 of them use manual toothbrushes and 15 of them use electric toothbrushes) participated in the study. 12 teeth of each individual, including upper and lower anteriors, were examined. The researchers supplied the volunteers with a manual toothbrush (Oral-B toothbrush Pro Expert Complete, Procter&Gamble, USA), an electronic toothbrush with replacement head (Oral-B Cross Action toothbrush replacement head, Procter&Gamble, USA), and a toothpaste (Oral-B Professional Toothpaste and Enamel Pro Repair Toothpaste, Procter&Gamble, USA).

Changing the Type of Toothbrush The first group (Group 1) includes volunteers who used to use manual toothbrushes and started to use an electric toothbrush for 1 month with the same daily brushing routine. The second group (Group 2) includes volunteers who used to use an electric toothbrush and started to use a manual toothbrush for 1 month with the same daily brushing routines.

Plaque and gingival index measurements Following the clinical intraoral examination of the volunteers in both groups, plaque and gingival index measurements were performed 5 hours after brushing. Regarding the plaque detection, a special 3-tone plaque staining product, Tri Plaque ID gel (GC Corp., Tokyo, Japan), was used to demonstrate the quantity and quality of the plaques on teeth' surfaces. The staining gel was applied onto buccal surfaces of upper and lower anterior teeth. The plaque and gingival indexes were both evaluated initially, 1 week, and 1 month after the toothbrush changes. The plaque index was evaluated according to Quigley and Hein's Plaque Index criteria. The gingival index was evaluated through Sillness & Löe Gingival Index and was scored clinically on visual inspection, digitally on dental photographs and digital imaging systems.

Quigley ve Hein Plaque Index 0 -> No plaque 1 -> Flecks of stain of the gingival margin 2 -> Definitive line of plaque on gingival margin 3 -> Gingival third of surface 4 -> Two-thirds of surface 5 -> Greater then 2/3rd of the surface Sillness & Löe Gingival Index 0 -> Healthy gingiva 1 -> Slight change in color and mild inflammation, no bleeding 2 -> Redness, moderate inflammation, bleeding on probing/pressure 3 -> Marked redness, severe inflammation, spontaneous bleeding Monitorization with intraoral dental photography The stained and unstained photographs of the teeth were taken initially, one week, and one month after the toothbrush changes. A camera (Nikon D7100), a macro lens (Nikon, 105mm VR macro lens), and a TTL dual macro flashlight (Meike MK-MT24N) was used for the DSLR photography. The camera parameters were set to ISO 400, diaphragm f/25, and shutter speed 1/125. A mobile dental photography device, Smile Lite MDP, was also used in combination with a smart phone (iPhone 12 Mini, Apple Inc, CA, USA) as an alternative photography technique. CP filter was used for all the photographs taken with Smart Lite MDP. The photographs with and without CP were taken without calibrating the white balance (WB) in auto white balance (AWB) mode. Additionally, a led curing unit D-Light Pro was used in detection mode in combination with the DSLR camera to enhance the visualization of the stained plaque. ISO was set at 1600 and diaphragm f/11 for photography with the D-Light Pro. The quantity of the plaque on tooth surfaces was scored through the photographic analysis.

Monitorization with digital imaging systems The stained and unstained measurements were performed initially, one week, and one month after the toothbrush changes by using FluoreCam and iTero Flex devices. After the plaque was stained, it was distinguished from healthy enamel tissue in terms of both color and fluorescence properties. FluoreCam device was used as one of the methods to determine the amount of dental plaque visually and numerically in this study. The stained plaque areas were automatically marked and recorded in the FluoreCam software, simultaneously with the visualization of fluorescence images of upper and lower anterior teeth on the screen. Size and intensity values of stained plaque were obtained from FluoreCam software. Size values represent the area of the plaque, meanwhile intensity values demonstrate the amount of mineral loss and were always represented as a negative number. Decreasing values in intensity (e.g., from -15 to -10) signify that the lesion (mineral content) had slightly improved.

The images of the anterior teeth were also taken by using a real-time intraoral scanner, iTero Element Flex (AlignTech, Carlstadt, USA) to digitalize and distinguish the plaque dye to provide clear 3D images and better visual assessment.

Plaque measurements and gingival index scores at initial, one week, and one month after the toothbrush change; for Group 1 and Group 2 were evaluated statistically using Mann Whitney U test. Additionally, the images obtained by the FluoreCam device were compared on the system software and evaluated statistically using Mann Whitney U and Wilcoxon tests.

ELIGIBILITY:
Inclusion Criteria:

* using manual or electric toothbrush for at least 2 years

Exclusion Criteria:

* systemic disease,
* restoration or caries in anterior teeth

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Plaque index | 1 week
  Plaque was evaluated according to Quigley and Hein's Plaque Index criteria
Gingival index | 1 week
  Gingival index was evaluated through Sillness&Löe Gingival Index
Fluorescence assesment | 1 week
  FluoreCam device is based on fluorescence technology. After dental plaque is stained, it is distinguished from healthy enamel tissue in terms of both color and fluorescence properties. FluoreCam system's software determines the amount of dental plaque visually and quantitatively. The stained plaque areas were automatically marked and recorded in the FluoreCam software, simultaneously with the visualization of fluorescence images of upper and lower anterior teeth on the screen. Size and intesity values of stained plaque were obtained from FluoreCam software.
intraoral dental photography | 1 week
  dental plaque was evaluated using a digital camera and mobile dental photography device and scored according to Quigley and Hein's Plaque Index
intraoral scanner | 1 week
  plaque was evaluated visually using iTero Flex intraoral scanner

SECONDARY OUTCOMES:
Plaque index | 1 month
  Plaque was evaluated according to Quigley and Hein's Plaque Index criteria
Gingival index | 1 month
  Gingival index was evaluated through Sillness&Löe Gingival Index
Fluorescence assesment | 1 month
  FluoreCam device is based on fluorescence technology. After dental plaque is stained, it is distinguished from healthy enamel tissue in terms of both color and fluorescence properties. FluoreCam system's software determines the amount of dental plaque visually and quantitatively. The stained plaque areas were automatically marked and recorded in the FluoreCam software, simultaneously with the visualization of fluorescence images of upper and lower anterior teeth on the screen. Size and intesity values of stained plaque were obtained from FluoreCam software.
intraoral dental photography | 1 month
  dental plaque was evaluated using a digital camera and mobile dental photography device and scored according to Quigley and Hein's Plaque Index
intraoral scanner | 1 month
  plaque was evaluated visually using iTero Flex intraoral scanner

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Tağtekin, Prof. Dr., Study Director — Marmara University Faculty of Dentistry Department of Restorative Dentistry; Elif Alkan, Res. Asst., Principal Investigator — Marmara University Faculty of Dentistry Department of Restorative Dentistry; Ataberk Kayhan, Student, Study Chair — Marmara University Faculty of Dentistry
Locations (1):
- Marmara University Faculty of Dentistry, Istanbul, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data obtained from the study will be presented and published internationally
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after the article is published.
Access Criteria: After the article published, corresponding author will share the data when asked.

REFERENCES:
- [Background] QUIGLEY GA, HEIN JW. Comparative cleansing efficiency of manual and power brushing. J Am Dent Assoc. 1962 Jul;65:26-9. doi: 10.14219/jada.archive.1962.0184. No abstract available. PMID 14489483
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Abufarwa M, Noureldin A, Campbell PM, Buschang PH. Reliability and validity of FluoreCam for white-spot lesion detection: An in vitro study. J Investig Clin Dent. 2018 Feb;9(1). doi: 10.1111/jicd.12277. Epub 2017 Jun 20. PMID 28631885